CLINICAL TRIAL: NCT01196455
Title: Phase II Clinical Study of Capecitabine in Combination With Mitomycin C as First-Line Treatment in Patients With Metastatic Breast Cancer
Brief Title: Capecitabine and Mitomycin C in Treatment of Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Croatian Cooperative Group for Clinical Research in Oncology (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Prof. dr. sc. Eduard Vrdoljak, Clinical Hospital Split, Center of oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO18646
Record Dates: First submitted 2010-08-31; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-08

CONDITIONS: Breast Cancer; Metastasis
Keywords: Metastatic breast cancer patients
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine and Mitomycin C — * Capecitabine 1000 mg/m2 twice-daily, administered orally on day 1-14, every three weeks
  * Mitomycin C 8 mg/m2 i.v. bolus, on day 1, every three weeks
  Other Names: Capecitabine (Xeloda); Mitomycin C (Mutamycin)

SUMMARY:
This is an open-label, non-comparative efficacy and safety study of Capecitabine and Mitomycin C as first-line treatment in patients with previously untreated metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed breast cancer
* Metastatic breast cancer, having at least one target lesion according to the RECIST criteria. Bone metastases, leptomeningeal disease, ascites, pleural or pericardial effusions, inflammatory breast disease, lymphangitic spread or cystic lesions are not acceptable as target lesions. Target lesions must be ≥ 10 mm longest diameter measured in one dimension using spiral CT, or ≥ 20 mm longest diameter measured in one dimension using conventional techniques. In addition to the definitions pertaining to the target lesion(s) from the RECIST criteria above, the target lesion(s) must not have been previously irradiated (newly arising lesions in previously irradiated areas are acceptable).
* Age > 18 years
* Signed informed consent obtained prior to initiation of any study-specific procedures or treatment

Exclusion Criteria:

* Prior cytotoxic chemotherapy or active/passive immunotherapy for metastatic breast disease
* Prior usage of capecitabine or mitomycin as adjuvant or neoadjuvant treatment
* Life expectancy < 3 months
* Not-ambulatory or with an ECOG performance status > 1
* Insufficient hematological, renal and hepatic functions:
* hemoglobin < 8.0 g/dL
* absolute neutrophils count (ANC) < 1.5 x 109/L
* platelet count < 100 x 109/L
* serum creatinine > 1.25 x N*
* total bilirubin > 2.0 x N*
* ASAT and/or ALAT > 2.5 x N* (in case of liver metastases > 5 x N*)
* alkaline phosphatase > 2.5 x N* (in case of liver metastases > 5 x N*, in case of bone metastases > 10 x N*) *N = upper limit of standard range
* Severe renal impairment [creatinine clearance < 30 mL/min (calculated according to cockcroft and Gault)]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Response rate | average 5 years

SECONDARY OUTCOMES:
time to disease progression | average 5 years
overall survival | average 5 years
Toxicity | average 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vrdoljak, MD PhD, Principal Investigator — Clinical Hospital Split, Center of oncology, Croatia
Locations (1):
- Center of oncology, Split, Croatia